CLINICAL TRIAL: NCT06635733
Title: A Cluster Randomized Controlled Trial of the Pediatric Acute Care Education (PACE) Program Combining Adaptive E-Learning with In-Person Skills Practice in Tanzania
Brief Title: Enhancing Pediatric Acute Care Through Adaptive E-Learning and In-Person Skills Practice in Tanzania
Acronym: PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Catholic University of Health and Allied Sciences (Other); London School of Hygiene and Tropical Medicine (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Peter A Meaney, MD MPH, Clinical Professor, Pediatric Critical Care, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R21TW012612-01A1-2025; 1R21TW012612-01A1 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Newborn Resuscitation; Severe Malnutrition; Severe Malaria; Severe Pneumonia; Severe Dehydration; In-Service Training; Computer-Assisted Instruction; Simulation Training
Keywords: Pediatric acute care; Newborn resuscitation; Severe malnutrition in children; Severe malaria treatment; Severe dehydration management; Pediatric pneumonia care; In-person skills practice (ISP); Adaptive e-learning for healthcare providers; Clinical skills training in low-resource settings; Health provider education; Clinical champions; Tanzania healthcare providers; Pediatric emergency training; Blended learning in pediatric care; Refresher learning progress (RLP); Cluster randomized controlled trial (RCT); Rhapsode Capable™ platform; Skills assessment in pediatric care; Continuous professional development (CPD) for healthcare providers
MeSH Terms: conditions — Malnutrition; Malaria; Pneumonia; Dehydration; Child Nutrition Disorders; Cephalopelvic Disproportion | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study is a cluster randomized controlled trial (RCT) where healthcare providers are assigned to either the intervention group, which uses the Rhapsode Capable™ platform for in-person skills practice (ISP) scheduling, feedback, and assessment, or the control group, which follows paper-based ISP. Both groups receive the same Pediatric Acute Care Education (PACE) adaptive learning content, but the method of ISP differs between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Rhapsode Capable™ Platform) (Experimental): Participants (healthcare providers) in this group will receive the PACE adaptive learning modules and participate in In-Person Skills Practice (ISP) sessions facilitated by clinical champions. The ISP sessions will be managed using the Rhapsode Capable™ platform, which allows for scheduling, real-time performance feedback, and tracking of progress. The intervention is designed to enhance pediatric care competencies by blending adaptive e-learning with structured, feedback-driven skills practice.
  Interventions: Behavioral: Rhapsode Capable™ Platform (Intervention Group)
- Control Group (Paper-based ISP) (Active Comparator): Participants (healthcare providers) in this group will also receive the same PACE adaptive learning modules and participate in In-Person Skills Practice (ISP) sessions facilitated by clinical champions. However, ISP sessions will be conducted using paper-based assessments. Clinical champions will manually track performance, provide feedback, and schedule sessions using paper forms. The control group will not have access to real-time digital feedback or automated progress tracking.
  Interventions: Behavioral: Paper-based ISP (Control Group)

INTERVENTIONS:
Behavioral: Rhapsode Capable™ Platform (Intervention Group) — Participants in the intervention group will use the Rhapsode Capable™ platform to facilitate In-Person Skills Practice (ISP) sessions. The platform allows for scheduling ISP sessions, providing real-time performance feedback, and tracking progress. The platform integrates with the PACE adaptive learning modules, which cover pediatric acute care topics. The goal is to improve skills retention and performance in pediatric care through a blended learning approach.
  Arms: Intervention Group (Rhapsode Capable™ Platform)
Behavioral: Paper-based ISP (Control Group) — Participants in the control group will also receive In-Person Skills Practice (ISP) sessions facilitated by clinical champions, but without the use of the digital platform. The ISP sessions will be tracked and scheduled using paper-based assessments. Feedback will be provided verbally or manually, and progress will be documented using paper forms. Both groups will receive the same PACE adaptive learning modules, but the method of ISP implementation differs between the groups.
  Arms: Control Group (Paper-based ISP)

SUMMARY:
The goal of this clinical trial is to evaluate whether the integration of in-person skills practice (ISP) with an adaptive e-learning platform can improve refresher learning progress (RLP) among healthcare providers in pediatric care settings in Tanzania.

The main questions it aims to answer are:

Can healthcare providers who participate in ISP sessions facilitated by clinical champions achieve greater improvements in refresher learning progress (RLP)? Will providers in the intervention group demonstrate improved metacognition and practical skill performance compared to those in the control group? Researchers will compare healthcare providers using the ISP digital platform (Rhapsode Capable™) to providers using paper-based ISP to see if the digital platform results in significantly higher RLP and fewer skill-based errors.

Participants will:

Complete adaptive e-learning modules focused on pediatric care topics (e.g., newborn resuscitation, severe malnutrition).

Participate in ISP sessions where clinical champions provide feedback and assess performance.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled trial (RCT) aimed at assessing the effectiveness of integrating In-Person Skills Practice (ISP) sessions facilitated by clinical champions into the existing Pediatric Acute Care Education (PACE) adaptive e-learning program. The study is designed to evaluate whether this blended learning approach can enhance the refresher learning progress (RLP), improve practical clinical skills, and increase metacognition (conscious competence) among healthcare providers responsible for pediatric care in Tanzania.

Study Design:

The trial will randomize four healthcare centers into two groups: an intervention group where providers use the Rhapsode Capable™ platform for ISP and a control group where providers receive paper-based ISP. Both groups will receive the same core content from the PACE adaptive learning modules.

The intervention group will utilize the Rhapsode Capable™ digital platform for ISP, which provides scheduling, skill tracking, and real-time feedback on performance. The control group will follow a similar protocol, but feedback and skill tracking will be done manually using paper forms. Clinical champions will facilitate all ISP sessions in both groups, providing structured guidance, peer support, and real-time feedback.

This trial will use a mixed-methods approach, including quantitative assessments (learning progress scores, ISP scores) and qualitative data collection (Focus Group Discussions and In-Depth Interviews) to gather insights into the barriers and facilitators of ISP integration into the PACE program.

Study Procedures:

1. Intervention Group:

   Healthcare providers will complete core PACE adaptive e-learning modules, focusing on pediatric care topics like newborn resuscitation, severe malnutrition, severe malaria, and respiratory conditions.

   Providers will participate in ISP sessions facilitated by clinical champions using the Rhapsode Capable™ platform. These sessions will provide an opportunity for providers to practice critical clinical skills with real-time feedback and scoring.

   The platform will track provider progress, enabling personalized feedback based on performance, scheduling of future sessions, and consistency of practice.
2. Control Group:

Providers will complete the same core PACE adaptive e-learning modules. ISP sessions will be conducted using paper-based assessments facilitated by clinical champions. Feedback will be provided verbally during sessions, and scores will be recorded manually.

Quality Assurance Procedures:

To ensure data integrity and consistent delivery of the intervention, several quality assurance measures will be implemented:

Data Validation: Data entered into the Rhapsode Capable™ platform for the intervention group will undergo automated validation checks for consistency, range, and completeness. For the control group, the PACE coordinator will perform weekly reviews of paper forms and cross-check them against participant logs.

Site Monitoring: Clinical champions and the study coordinator will conduct regular site visits to monitor compliance with ISP protocols, data collection, and participant engagement.

Source Data Verification (SDV): Random checks of paper-based ISP assessments will be compared with original session records to verify accuracy and completeness.

Standard Operating Procedures (SOPs): The study will adhere to detailed SOPs for each aspect of the trial, including participant recruitment, ISP facilitation, data management, and reporting of adverse events.

Data Management:

Data Collection: Data will be collected via the Rhapsode Capable™ platform (for the intervention group) and manual paper forms (for the control group). All data will be transferred to the secure REDCap database for analysis.

Data Checks: A dedicated PACE coordinator will regularly perform data checks to compare ISP scores, ensure participant progression, and resolve any discrepancies in the dataset.

Data Dictionary: A detailed data dictionary will be maintained, outlining each variable, its source, coding system, and any range limits. This will include information about ISP performance scores, learning progress metrics, demographic data, and survey results.

Sample Size:

The trial will enroll 90 healthcare providers (45 in the intervention group and 45 in the control group). After accounting for a potential dropout rate of up to 10%, it is expected that 80 providers will complete the full study protocol. This sample size is calculated based on anticipated differences in the primary outcome (RLP) and allows for detection of significant differences between the two groups with a power of 80% at a significance level of 0.05.

Plan for Missing Data:

A comprehensive plan for managing missing data will be implemented:

Imputation Methods: Missing data will be addressed using multiple imputation techniques if the missing data exceeds 5%. In cases where data is missing completely at random (MCAR), a complete case analysis will be conducted.

Handling Data Inconsistency: Any inconsistent or out-of-range data will be flagged during weekly data checks and verified by clinical champions or the PACE coordinator.

Statistical Analysis:

The primary analysis will focus on comparing the median refresher learning progress (RLP) between the intervention and control groups. Statistical significance will be determined using the Wilcoxon rank-sum test to account for the non-parametric distribution of data. A two-sided alpha of 0.05 will be used for hypothesis testing.

The secondary analyses will include:

Changes in metacognition (conscious competence) using generalized estimating equations (GEE) to account for repeated measures over time.

ISP scores between intervention and control groups using mixed-effects linear regression models, adjusting for baseline ISP scores.

Trends in common errors observed during ISP sessions. The trial will also conduct an exploratory analysis of the qualitative data collected through Focus Group Discussions (FGDs) and In-Depth Interviews (IDIs). This data will be analyzed using thematic analysis, focusing on participant feedback regarding the ease of ISP integration, the perceived value of clinical champions, and any barriers encountered during the study.

Registry Information:

Registry Procedures: To maintain data accuracy and ensure consistent participant monitoring, the PACE program will include:

On-site Audits: Routine on-site audits will be conducted to verify data accuracy and adherence to ISP protocols.

Data Entry Audits: Manual data entry (for the control group) will be reviewed weekly by the PACE coordinator, and discrepancies will be addressed immediately.

Monitoring Plan: Weekly educator dashboard summaries will be provided to clinical champions, highlighting provider progress and any outstanding ISP tasks.

Ethical Considerations:

This study has been approved by the Institutional Review Boards (IRBs) of the Catholic University of Health and Allied Sciences (CUHAS), Stanford University, and London School of Hygiene and Tropical Medicine (LSHTM). Ethical concerns such as data confidentiality and informed consent have been thoroughly addressed, and all participants will be able to withdraw from the study at any point without penalty.

Conclusion:

The results of this study will provide critical insights into the effectiveness of integrating adaptive e-learning with in-person skills practice to improve pediatric care in low-resource settings. If successful, the findings could lead to the implementation of scalable, blended learning strategies to improve healthcare outcomes for children in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers actively involved in pediatric care at one of the selected healthcare centers.
* Completion of core Pediatric Acute Care Education (PACE) adaptive learning modules prior to study participation.
* Willingness to participate in In-Person Skills Practice (ISP) sessions.
* Ability to engage with either the Rhapsode Capable™ platform (intervention group) or paper-based ISP methods (control group).
* Minimum proficiency in written and spoken English.

Exclusion Criteria:

* Healthcare providers not involved in pediatric or newborn clinical care at the time of recruitment.
* Providers unable or unwilling to attend ISP sessions facilitated by clinical champions.
* Individuals with no prior engagement in the PACE program.
* Providers with significant technological barriers that prevent the use of the Rhapsode Capable™ platform (for the intervention group only).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Median Refresher Learning Progress (RLP) Among Providers | 16 (Pilot) or 32 (repilot) weeks from baseline to study completion. Each participant's progress will be tracked weekly throughout the 16/32-week intervention period.
  The percentage of refresher learning modules completed by healthcare providers with an initial learning progress (ILP) score of 95% or greater, who also complete at least one In-Person Skills Practice (ISP) session per month. The RLP will be measured as the progress in refresher module completion and adherence to ISP sessions, indicating the effectiveness of combining adaptive e-learning with in-person skills practice.

SECONDARY OUTCOMES:
Improvement in Metacognition (Conscious Competence) | Assessed at baseline, 16 weeks(pilot only), and 32 weeks (repilot only) after intervention start.
  The degree of improvement in metacognition will be assessed using Howell's metacognition categories, which include conscious competence, unconscious competence, conscious incompetence, and unconscious incompetence. Providers will be evaluated on their ability to accurately recognize their clinical skills and knowledge across these categories. The focus will be on shifts from unconscious incompetence and conscious incompetence to conscious competence and unconscious competence as providers progress through the intervention.
Total ISP Score Improvement | Assessed after each ISP session and summarized at 16 (pilot) or 32 (repilot) weeks after intervention start.
  The overall improvement in ISP (In-Person Skills Practice) performance scores. ISP sessions will be evaluated using structured observation forms, and improvements will be tracked across multiple pediatric clinical skills, such as newborn resuscitation and management of severe pediatric conditions. Scores will be based on specific skill proficiency and adherence to pediatric care protocols.
Reduction in Common ISP Errors | Errors tracked throughout ISP sessions over the 16 or 32-week intervention period.
  The frequency and type of common errors observed during ISP sessions. Clinical champions will document provider errors during ISP sessions, and the data will be analyzed to determine whether the intervention reduces the number of skill-based errors over time compared to the control group.
Proportion of Healthy Providers (HPs) | Assessed monthly and summarized at 16 or 32 weeks after intervention start.
  The proportion of healthcare providers who achieve and maintain an Initial Learning Progress (ILP) of 95% or greater and participate in at least one ISP session per month. A "healthy provider" is defined as one who consistently meets these criteria over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Meaney, MD MPH, Principal Investigator — Stanford University; Adolfine Hokororo, MD, Principal Investigator — Catholic University of Health and Allied Sciences
Locations (1):
- Catholic University of Health and Allied Sciences, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The study will share individual participant data (IPD) that underlie the results reported in publications arising from this clinical trial. This will include de-identified data for all variables used in analyses, such as demographic data, learning progress metrics, and ISP scores. The shared data will be provided with supporting documentation to ensure transparency and reproducibility.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be made available starting 6 months after publication of the primary study results and will be available for a period of 5 years from that date.
Access Criteria: Access to the shared IPD will be granted to researchers who submit a formal request with a scientifically sound proposal for secondary analyses. Proposals will be reviewed by the study team members, data access committee, and access will be granted via a secure data-sharing platform. Researchers will be required to sign a data use agreement ensuring the protection of participant confidentiality and adherence to ethical use of the data.